CLINICAL TRIAL: NCT06028646
Title: Dynamic Airway CT is Diagnostic for Tracheomalacia in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-01279
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Tracheomalacia
Keywords: Tracheomalacia in Children
MeSH Terms: conditions — Tracheomalacia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dynamic Airway CT scan (DA-CT) (Experimental): All participants will have a DA-CT scan after flexible bronchoscopy has been performed.
  Interventions: Device: Dynamic Airway CT scan (DA-CT)

INTERVENTIONS:
Device: Dynamic Airway CT scan (DA-CT) — Patient will be asked to perform movements during the scan.

SUMMARY:
The purpose of this pilot interventional study is to evaluate the use of Dynamic Airway Computed Tomography (DA-CT) for diagnosis of tracheomalacia in children 0-18 years for whom flexible bronchoscopy has been performed. The primary aims are to evaluate the diagnostic accuracy, image quality, and radiation exposure of DA-CT as a potential noninvasive alternative to the gold standard of flexible bronchoscopy in the diagnosis of tracheomalacia. The results from this pilot study will help to estimate sample size for a larger-scale study with more precise estimates of DA-CT diagnostic potential.

ELIGIBILITY:
Inclusion Criteria:

* Participants 0-18 years old, with
* Clinically indicated flexible bronchoscopy has been performed

Exclusion Criteria:

* Pregnancy or breastfeeding
* Unable to undergo CT scanning without sedation
* Patients with tracheostomy

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Severity of dynamic narrowing on Flexible Bronchoscopy | Through study completion, an average of 1 year
  Video recordings and images will be deidentified and reviewed by pediatric pulmonologists and scores averaged.
  Severity of dynamic narrowing will be classified as follows: mild: 50%-74%, moderate: 75%-89%, severe: >90%.
Severity of Maximal Airway Change (MAC) on DA-CT | Through study completion, an average of 1 year
  Severity of MAC will be classified as follows: mild: 33%-49%, moderate: 50%-66%, severe: >67%.
  This outcome will be measured using the following equation:
  MAC = tracheal cross-sectional (CSA) at narrowed segment in inspiration/CSA of trachea at thoracic inlet in inspiration
Severity of Excessive dynamic airway collapse (EDAC) on DA-CT | Through study completion, an average of 1 year
  Severity of EDAC will be classified as follows: mild: 50%-74%, moderate: 75%-89%, severe: >90%.
  This outcome will be measured using the following equation:
  EDAC = CSA at airway segment in expiration/CSA at same location in inspiration

SECONDARY OUTCOMES:
Contrast-to-noise-ratio (CNR) of DA-CT scanners | Through study completion, an average of 1 year
  This outcome will be measured using the following equation:
  CNR = (mean Hounsfield Units (HU) in the artery regions of interest (ROI) - mean HU in the tracheal air column ROI) / image noise inside the trachea.
Qualitative Analysis of DA-CT Image Quality based on 5-point Likert scale | Through study completion, an average of 1 year
  5-point Likert scale will be used as follows: (1) Very Poor, (2) Poor, (3) Fair, (4) Good, (5) Excellent
Qualitative Analysis of DA-CT image noise based on 5-point Likert scale | Through study completion, an average of 1 year
  5-point Likert scale will be used as follows: (1) Very Poor, (2) Poor, (3) Fair, (4) Good, (5) Excellent
Qualitative Analysis of DA-CT delineation of large airways based on 5-point Likert scale | Through study completion, an average of 1 year
  5-point Likert scale will be used as follows: (1) Very Poor, (2) Poor, (3) Fair, (4) Good, (5) Excellent
Qualitative Analysis of DA-CT delineation of small airways based on 5-point Likert scale | Through study completion, an average of 1 year
  5-point Likert scale will be used as follows: (1) Very Poor, (2) Poor, (3) Fair, (4) Good, (5) Excellent
Qualitative Analysis of DA-CT noise texture based on 5-point Likert scale | Through study completion, an average of 1 year
  5-point Likert scale will be used as follows: (1) Very Poor, (2) Poor, (3) Fair, (4) Good, (5) Excellent
Radiation exposure of DA-CT scanners | Through study completion, an average of 1 year
  The effective dose (in mSv) will be automatically calculated with tissue weighting factors

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Muise, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Fink Children's Ambulatory Center/Hassenfeld Children's Center, New York, New York
  - Tisch Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Eleanor.Muise@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Eleanor.Muise@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.